CLINICAL TRIAL: NCT04633538
Title: Evaluation of a New 6 Minute Walk Test Smartphone App in Patients With Pulmonary Hypertension (The 6-APP Study)
Brief Title: Evaluation of a New 6 Minute Walk Test Smartphone App in Patients With Pulmonary Hypertension
Acronym: 6-APP
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Elizabeth Orchard, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: PID13040
Record Dates: First submitted 2020-08-26; First posted 2020-11-18 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 6MWT app group: Patients who received the 6MWT app and performed tests at the clinic and in the community using the app
  Interventions: Device: 6MWT smartphone app

INTERVENTIONS:
Device: 6MWT smartphone app — Use of smartphone app to measure 6 minute walk test (6MWT)

SUMMARY:
Comparison of standard 6 minute walk test with 6 minute walk test smartphone app.

DETAILED DESCRIPTION:
Pulmonary Arterial Hypertension (PAH) is a progressive illness that; if not diagnosed early or left untreated, can be a severe life limiting condition . It is a chronic disease of the pulmonary vasculature, with vascular proliferation and remodelling of the small pulmonary arteries leading to a progressive increase in pulmonary vascular resistance (PVR). This can ultimately lead to right heart failure and premature death . The predominant symptom of PAH is dyspnoea on exertion, with a decrease in exercise capacity, and most patients present with this symptom .

PAH is an uncommon condition, affecting about 6000 patients in the United Kingdom , and due to its rarity, the NHS commissions 7 centres to care for patients with PAH. Oxford University Hospital NHS Foundation Trust works closely with the Royal Brompton Hospital to provide care for patients with PAH in Oxfordshire and the surrounding region.

The six-minute walk test (6MWT) is a standard method for measuring exercise capacity in patients with cardiopulmonary disease such as PAH. The 6MWT measures how far a patient can walk in 6 minutes. Walking is an activity performed every day, by most patients except for those most severely limited. By assessing patients' ability to exercise, the 6MWT provides a global assessment of respiratory, cardiovascular, neuromuscular and cognitive function. The 6MWT does not differentiate what limits the patient, nor does it assess maximal exercise capacity. Instead, the 6MWT allows the patient to exercise at a daily functional level, and is a useful tool for assessing changes after a therapeutic intervention, and correlates with a subjective improvement in dyspnoea .

In PAH the 6MWT is used to evaluate patients' response to treatment, with an increase in 6MWT distance of greater than 42m being considered a clinically significant improvement . Furthermore, change in 6MWT distance correlates with VO2 max (maximum rate of oxygen consumption measured during exercise), NYHA class (classification of patients' daily limitation) and mortality in PAH patients, providing an objective assessment of disease progression, prognosis and response to treatment. It is a universally accepted test as it is safe and easily performed by the patient.

The 6MWT has become the primary end-point for many trials, and as a surrogate invalidated survival outcome for all placebo controlled trials of PAH therapy . It is used by regulatory bodies to determine whether a treatment should be approved. However, there is much discrepancy between whether it is the total distance walked at baseline prior to treatment, a decrease in total distance walked over time or a percentage increase in walking distance that correlates best with survival outcome. The investigators hypothesize that it is all 3 of these measures, and that having a validated and more reproducible 6MWT would help assess patients and guide treatment strategies better.

The test is usually performed in hospital, by walking along a hospital corridor, where many factors on the day of the test can affect patients' performance, including tiredness, unfamiliarity with the environment or anxiety. The test typically requires 2 physiologists to monitor the distance walked by the patient, their oxygen saturations by pulse oximetry, and to record symptoms felt during the test. To improve the assessment of a patient's exercise capacity using a 6MWT, the investigators hypothesize that the test would reflect more the patient's functional status, if it were undertaken prior to the hospital outpatient appointment. The investigators have designed a mobile-phone "app" that allows patients to perform the 6MWT within the patient's home environment. This is felt to be more appealing to the patients, and would reduce the time spent in hospital on the day of their outpatient appointment.

The 6MWT app is categorised as a mobile-health (m-health) system, a form of telehealth whereby healthcare is delivered at a distance using smartphones. By utilizing biometric collection devices such as a pulse oximeter monitor with Bluetooth capability, m-health can be used to measure the oxygen saturation levels in the blood from patients, and transmit them to a secure server, allowing them to be reviewed by cardiologists and other healthcare professionals.

The evidence-base for m-health as a tool for assessing physical fitness is increasingly established. This new approach not only offers the opportunity for reliable collection of data, but provides the infrastructure to do this at scale and will allow decisions on patients' health to be based on more frequent and more accurate information.

There are no known risks to undertaking a 6MWT in the community as walking is an activity of daily living, and all patients are encouraged to walk daily.

The population to be studied will be those with PAH who are currently assessed with a 6MWT. Once the app has been validated, patients with any type of cardiorespiratory disease who are assessed with a 6MWT could use the app, for example patients with chronic obstructive airways disease, heart failure, renal failure, and pre-transplantation work up.

The 6MWT results form part of the NHS data set collected by NHS England for patients with PAH, and it would be beneficial to have a more reproducible assessment, whose results could be compared between the 7 centres providing care for these patients. At present, there is much variability in how 6MWTs are performed between units, and the app would reduce this variability.

The 6MWT has been undertaken at the John Radcliffe hospital for 5 years and the investigators will also retrospectively analyse the data from the 6MWT that have previously been undertaken. The data on patients will be pseudo-anonymised, i.e. no personal information like name, surname or address, will be used, but the investigators will keep date of birth, gender, diagnosis, dates and results of the 6MWT, date and causes of death. As part of the clinical care team, reviewing the data is part of the normal standard of care for patients with PHT. The data is collected on the Solus cardiac reporting system and can be extracted from this database. The data will be pseudo-anonymised by the Principle Investigator for analysis, and then shared with the wider research team. The data will be analysed to look at distance walked, and change in oxygen saturation and heart rate during the test. The investigators will analyse the data over time, to look for changes in these parameters and correlate these with outcome data, i.e. mortality.

The study aims at demonstrating that patients are able and willing to use the app for the 6MWT and the measurements obtained by the app are comparable to the ones obtained in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above
* Diagnosed with PAH who are able to undertake 6MWT off-oxygen
* Being of PAH group 1 or 4
* Participant owns a compatible smartphone (Android or iPhone) and is able to use it.

Exclusion Criteria:

* Long term oxygen therapy
* Cognitive impairments
* Rheumatological diseases that limit the measurement of finger Oxygen saturations
* PAH groups 2, 3 or 5
* Cannot use a smartphone
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing follow up in the PAH clinic will be eligible for participation. They will be approached by a member of the clinical team for consideration and recruited. We will recruit 30 compliant patients to enrol in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Orchard, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agarwal R, Gomberg-Maitland M. Current therapeutics and practical management strategies for pulmonary arterial hypertension. Am Heart J. 2011 Aug;162(2):201-13. doi: 10.1016/j.ahj.2011.05.012. Epub 2011 Jul 13. PMID 21835279
- [Background] Galie N, Brundage BH, Ghofrani HA, Oudiz RJ, Simonneau G, Safdar Z, Shapiro S, White RJ, Chan M, Beardsworth A, Frumkin L, Barst RJ; Pulmonary Arterial Hypertension and Response to Tadalafil (PHIRST) Study Group. Tadalafil therapy for pulmonary arterial hypertension. Circulation. 2009 Jun 9;119(22):2894-903. doi: 10.1161/CIRCULATIONAHA.108.839274. Epub 2009 May 26. PMID 19470885
- [Background] Tan MP, Bansal SK, Wynn NN, Umerov M, Gillham A, Henderson A, Hildreth A, Junejo S. Long term survival of patients with raised pulmonary arterial systolic pressure utilizing echocardiography-a five-year prospective study. J Geriatr Cardiol. 2012 Dec;9(4):328-35. doi: 10.3724/SP.J.1263.2012.06191. PMID 23341836
- [Background] Gabler NB, French B, Strom BL, Palevsky HI, Taichman DB, Kawut SM, Halpern SD. Validation of 6-minute walk distance as a surrogate end point in pulmonary arterial hypertension trials. Circulation. 2012 Jul 17;126(3):349-56. doi: 10.1161/CIRCULATIONAHA.112.105890. Epub 2012 Jun 13. PMID 22696079
- [Background] Mathai SC, Puhan MA, Lam D, Wise RA. The minimal important difference in the 6-minute walk test for patients with pulmonary arterial hypertension. Am J Respir Crit Care Med. 2012 Sep 1;186(5):428-33. doi: 10.1164/rccm.201203-0480OC. Epub 2012 Jun 21. PMID 22723290
- [Background] Miyamoto S, Nagaya N, Satoh T, Kyotani S, Sakamaki F, Fujita M, Nakanishi N, Miyatake K. Clinical correlates and prognostic significance of six-minute walk test in patients with primary pulmonary hypertension. Comparison with cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):487-92. doi: 10.1164/ajrccm.161.2.9906015. PMID 10673190
- [Background] Barst RJ, Rubin LJ, Long WA, McGoon MD, Rich S, Badesch DB, Groves BM, Tapson VF, Bourge RC, Brundage BH, Koerner SK, Langleben D, Keller CA, Murali S, Uretsky BF, Clayton LM, Jobsis MM, Blackburn SD, Shortino D, Crow JW; Primary Pulmonary Hypertension Study Group. A comparison of continuous intravenous epoprostenol (prostacyclin) with conventional therapy for primary pulmonary hypertension. N Engl J Med. 1996 Feb 1;334(5):296-301. doi: 10.1056/NEJM199602013340504. PMID 8532025
- [Derived] Salvi D, Poffley E, Tarassenko L, Orchard E. App-Based Versus Standard Six-Minute Walk Test in Pulmonary Hypertension: Mixed Methods Study. JMIR Mhealth Uhealth. 2021 Jun 7;9(6):e22748. doi: 10.2196/22748. PMID 34096876

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 6MWT App Group
Started | 30
Completed | 25
Not Completed | 5
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: We approached 33 patients; of these, 30 were eligible and consented to participate. Five patients withdrew from the study (3 were lost to follow-up, 1 died, and 1 considered the study not to be relevant any longer).
Arm/Group | 6MWT App Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 50 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Perform App-based Home 6MWT
Description: Percentage of participants who perform app-based home 6MWT.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 6MWT App Group
Number analyzed (Participants) | 30
Participants | 30

2. Secondary Outcome: Difference in Walked Distance Between 6MWT Test at the Clinic as Measured by Physiologists and the App in Indoor Mode
Description: Comparison of the indoor app-based 6MWD against simultaneous clinic 6MWD: mean and standard deviation of the difference in distance as measured by physiologists and the app. Differences at 3 time points (start, month 3 and month 6) are lumped together in the calculation of the statistics (mean and standard deviation).
Time Frame: At start, at month 3 and at month 6.
Population: 6MWT distances differences between conventional 6MWT in clinic, and using the app in indoor mode, simultaneously
Measure: Mean (Standard Deviation); unit: metre
Units Other Than Participants: Pairs of 6MWT distances
Groups:
- 6MWT App Group: Patients who performed tests at the clinic using the app simultaneously
Arm/Group | 6MWT App Group
Number analyzed (Participants) | 29
Number analyzed (Pairs of 6MWT distances) | 70
metre | 14.6 (75.48)

3. Secondary Outcome: Difference in Walked Distance Between 6MWT Test as Measured by Physiologists at the Clinic and App in Outdoor Mode at the Community
Description: Comparison of pairs of 6MWT distance estimates where one is the result of an observation done by a physiologist in a clinic (start, month 3 and month 6) and the other is measured by the app during an outdoor test performed within 7 days of the physiologist's observation. Measurements at 3 time points (start, month 3 and month 6) are lumped together in the calculation of the statistics (mean and standard deviation).
Time Frame: Clinic tests at start, at month 3, at month 6. Community tests undertaken within 7 days of clinic test.
Population: Difference of 6MWT distances, between conventional 6MWT in clinic, and using the app in outdoor mode in the community, within 7 days from clinic 6MWT
Measure: Mean (Standard Deviation); unit: metre
Units Other Than Participants: Pairs of 6MWT distances
Arm/Group | 6MWT App Group
Number analyzed (Participants) | 22
Number analyzed (Pairs of 6MWT distances) | 69
metre | 2.45 (47.0)

4. Secondary Outcome: Test-Retest Reliability of Community-Based 6MWT
Description: Intraclass correlation of app-base tests in outdoor mode in the community, measured over pairs of outdoor tests performed by the same patient no more than 7 days apart.
Time Frame: 6MWT in the community, at the patient's discretion (recommended once/month), over 6 months
Population: Pairs of outdoor tests performed by the same patient no more than 7 days apart
Measure: Number; unit: ICC
Units Other Than Participants: Pairs of 6MWT distances
Groups:
- 6MWT App Group: Patients who performed 6MWT in the community using the app, with at least 2 community 6MWTs within 7 days.
Arm/Group | 6MWT App Group
Number analyzed (Participants) | 10
Number analyzed (Pairs of 6MWT distances) | 89
ICC | 0.91

5. Secondary Outcome: Compliance to Monitoring Regime in the Community
Description: Percentage of patients who performed at least 1 app-based 6MWT in the community per month
Time Frame: At month 6
Measure: Count of Participants; unit: Participants
Groups:
- 6MWT App Group: Patients who received the 6MWT app and performed tests at the clinic and in the community using the app. Only patients who completed the study.
Arm/Group | 6MWT App Group
Number analyzed (Participants) | 25
Participants | 12

ADVERSE EVENTS:
Time Frame: 1 year
Description: 1 patient died
Arm/Group | 6MWT App Group
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT04633538/Prot_SAP_000.pdf